CLINICAL TRIAL: NCT04924725
Title: National Taiwan University Hospital
Brief Title: Prospective Comparison of Diagnostic Accuracy Between Contrast-enhanced Harmonic and Conventional EUS-guided Fine-needle Biopsy in Solid Pancreatic Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 201810024RINC
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-01

CONDITIONS: Pancreatic Solid Lesions

STUDY DESIGN:
Intervention Model Description: The samples in each group will be sent for rapid onsite cytology evaluation (ROSE) and pathology evaluation. If diagnosis could be made after ROSE, the procedure will be stopped. Otherwise, the FNB with be repeated for at most six times in each group. In conventional group, if the diagnosis could be made within three times of FNB, we will inject Sonazoid and record the enhance pattern of the pancreatic lesion. If the diagnosis still undetermined, the patient will receive CEH-EUS-guided FNB as cross-over test.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEH-EUS-guided FNB group (Experimental): In CEH-EUS-guided FNB group, needle puncture directly to the enhancing area 15-20 times without passing to the non-enhancing area under CEH mode was performed.
  Interventions: Procedure: Endoscopic ultrasound-guided fine needle biopsy
- Conventional-EUS-guided FNB with fanning technique group (Active Comparator): In conventional-EUS-guided FNB with fanning technique group, the needle was positioned at four different areas within the mass and then moved back and forth four times in each area to procure tissue (4 × 4).
  Interventions: Procedure: Endoscopic ultrasound-guided fine needle biopsy

INTERVENTIONS:
Procedure: Endoscopic ultrasound-guided fine needle biopsy — Endoscopic ultrasound-guided fine-needle biopsy is used to collect biopsy samples from solid pancreatic lesions throughout the digestive tract and is useful in diagnosing solid pancreatic lesions

SUMMARY:
Endoscopic ultrasonography (EUS)-guided fine-needle aspiration/biopsy (FNA/B) is used to collect biopsy samples from many organs throughout the digestive tract and is useful in diagnosing solid pancreatic lesions (SPLs). The reported diagnostic accuracy of EUS-FNA for SPLs is 85-89.4%, the sensitivity is 82-94.7%, and the specificity is 100%. One randomized controlled trial reported that the fanning technique of FNA was superior to the standard approach because fewer passes were required to establish the diagnosis. However, in many cases, like SPLs with the presence of fibrosis and necrosis background, four or more needle passes are still needed to obtain sufficient biopsy samples. There is a potential risk of tumor seeding associated with multiple needle punctures. Therefore, it is important to minimize the number of needle passes.

Contrast-enhanced harmonic EUS (CEH-EUS) using sonazoid (Daiichi-Sankyo, Tokyo, Japan) is useful to visualize parenchymal perfusion in the pancreas and characterize of SPLs. Because the necrotic or fibrotic area within the SPLs were appeared as non-enhanced area, CEH-EUS could help us to avoid puncture the non-enhancing area hence increased the diagnostic accuracy. Katana et al. reported that conventional EUS-FNA has lower sensitivity (72.9%) for pancreatic adenocarcinoma with non-enhanced areas compared to with enhanced areas (94.3%) on CEH-EUS. Therefore, it would be difficult to obtain sufficient biopsy samples through unenhanced areas of SPLs.

DETAILED DESCRIPTION:
According to the study result by Katana et al., fanning technique in SPLs with avascular areas had a negative impact on diagnostic accuracy of FNA. Because of the retrospective basis of their study, a prospective study is warranted to answer whether CEH-EUS-guided FNA/B is superior to conventional EUS-guided FNA/B with fanning technique in SPLs. The main objective of this randomized trial therefore was to determine whether CEH-EUS-guided sampling to avoid non-enhanced areas within a mass lesion result in more rapid diagnosis requiring fewer FNA/B passes than the conventional EUS-guided FNA/B with fanning needle throughout the mass is targeted.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 20years
* Referred for EUS-guided tissue acquisition for solid pancreatic lesions
* The size of the lesion greater than 1cm in the largest diameter

Exclusion Criteria:

* Patients with coagulopathy or altered anatomy
* Contraindications for conscious sedation
* Pregnancy
* Patients cannot provide informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Total number of passes required to establish a diagnosis | 1 day
  The samples in each group will be sent for ROSE and pathology evaluation. If diagnosis could be made after ROSE, the procedure will be stopped. Otherwise, the FNB with be repeated for at most six times in each group.

SECONDARY OUTCOMES:
Diagnostic accuracy rate | 3 months
Overall complication rate | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuo YT, Chu YL, Wong WF, Han ML, Chen CC, Jan IS, Cheng WC, Shun CT, Tsai MC, Cheng TY, Wang HP. Randomized trial of contrast-enhanced harmonic guidance versus fanning technique for EUS-guided fine-needle biopsy sampling of solid pancreatic lesions. Gastrointest Endosc. 2023 Apr;97(4):732-740. doi: 10.1016/j.gie.2022.12.004. Epub 2022 Dec 9. PMID 36509113